CLINICAL TRIAL: NCT03005717
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of LIPO-202 (Salmeterol Xinafoate for Injection) for the Reduction of Submental Subcutaneous Fat
Brief Title: Study to Evaluate the Safety and Efficacy of LIPO-202 for the Reduction of Submental Subcutaneous Fat
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neothetics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LIPO-202-CL-31
Record Dates: First submitted 2016-12-21; First posted 2016-12-29 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Submental Fat
Keywords: submental; Salmeterol Xinafoate; LIPO-202; bulge
MeSH Terms: interventions — Salmeterol Xinafoate; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active High (Experimental): Drug: LIPO 202 (Salmeterol Xinafoate for Injection), 0.2 mcg SX/mL Total Weekly Dose: up to 3.0 mcg SX
  Interventions: Drug: LIPO-202
- Active Low (Experimental): Drug: LIPO 202 (Salmeterol Xinafoate for Injection), 0.02 mcg SX/mL Total Weekly Dose: up to 0.3 mcg SX
  Interventions: Drug: LIPO-202
- Placebo (Placebo Comparator): Placebo for LIPO 202 (Salmeterol Xinafoate for Injection)
  Interventions: Drug: Placebo for LIPO-202

INTERVENTIONS:
Drug: LIPO-202
  Other Names: Salmeterol Xinafoate for Injection
  Arms: Active High; Active Low
Drug: Placebo for LIPO-202 — Lyophile manufactured to mimic LIPO-202 lyophile.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Study LIPO-202-CL-31 is a multi center, randomized, double-blind, placebo-controlled study to evaluate the safety and efficacy of two different doses of LIPO-202 versus placebo on submental bulging due to subcutaneous fat. Approximately 150 participants of either gender who have a "Moderate Bulge" or "Large Bulge" in the submental fat (on Patient-Reported Submental Bulging Scale [PR-SBS] and Clinician-Reported Submental Bulging Scale [CR-SBS]) will be recruited for this study.

DETAILED DESCRIPTION:
Potential subjects will present and complete the Screening Visit. All qualifying subjects will be randomized to one of three treatment groups and treated with up to 30 subcutaneous injections of the assigned study drug into submental fat, once a week for 8 weeks. Upon completion of treatment visits, subject will return to the clinic for a follow-up visit and end of study visit, one and four weeks after the last treatment. The number and pattern of injections will be based on the area (cm x cm) of submental fat at baseline. At each visit the subjects will also undergo an examination of the treatment area, collection of vital signs and questioning about possible adverse events (AEs).

The study consists of 11 visits: a Screening Visit, eight Treatment Visits, a Follow up Visit and an End of Study Visit.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or non-pregnant females;
2. Capable of providing written, informed consent; and ,
3. Have submental bulging that is evaluated by the Investigator as "Moderate" or "Large".

Exclusion Criteria:

1. History of prior treatment to reduce submental bulging;
2. History of derm fillers, chemical peels, or laser or radio frequency procedures in the neck/chin area within 12 months of screening;
3. History of botulinum toxin in the neck/chin area within 6 months of screening;
4. Any skin conditions (including, but not limited to: skin infections, psoriasis, eczema, keloids, tattoos or hypertrophic or tethered scars) or history of trauma in the treatment area that may affect study procedures;
5. A score of 4 (Extreme Laxity) on the Skin Laxity Assessment Scale at Visit 1 (Screening);
6. Any known hypersensitivity to the study drug and/or any of the components;
7. Prior or current enrollment in any Lithera/Neothetics sponsored LIPO-102/LIPO-202 study;
8. Concurrently enrolled in another investigational drug or device study or used any experimental or investigational drug or device within 30 days of screening;
9. Female subject who is pregnant or lactating;
10. Any medical condition that in the opinion of the Investigator might complicate study procedures or assessments or jeopardize the subject's safety, including, but not limited to:

    1. any bleeding or connective tissue disorders;
    2. any clinically significant kidney or liver disease;
    3. any untreated thyroid disease;
    4. asthma, COPD, diabetes (Type I and II) or cardiovascular disease
    5. history of major surgery within 30 days prior to randomization, or planned surgery during the study period;
11. Used drugs with anticoagulant activity (including aspirin) within 14 days prior to randomization, β adrenergic receptor agonists or blockers, strong CYP3A inhibitors, or nonpotassium sparing diuretics (e.g., loop or thiazide diuretics) within 28 days prior to randomization;
12. Used tricyclic antidepressants or monoamine oxidase inhibitor medications within 14 days prior to randomization;
13. Unlikely or unable to adhere to the study visit schedule or comply with protocol procedures.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-06-02 (Actual)

PRIMARY OUTCOMES:
Safety as measured by number of subjects with adverse events. | 12 weeks (Baseline through 4 weeks post last dose)
Safety as measured by the number of subjects with abnormal post baseline shifts in laboratory results. | 12 weeks (Baseline through 4 weeks post last dose)
Change from baseline in the patient reported submental bulging scale. | 12 weeks (Baseline through 4 weeks post last dose)
  The self-rating scale is 5-point scale that the subject evaluates their submental fat.
Change from baseline in the clinician reported submental bulging scale | 12 weeks (Baseline through 4 weeks post last dose)
  The clinician scale is 5-point rating scale in which the clinician evaluates the subject's submental fat.
Change in submental fat thickness measured with calipers (mm). | 12 weeks (Baseline through 4 weeks post last dose)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Piacquadio, MD, Study Chair — Consultant, Therapeutics, Inc.
Locations (11):
- United States (11):
  - Clinical Testing of Beverly Hills, Beverly Hills, California
  - Ablon Skin Institute And Research Center, Manhattan Beach, California
  - AboutSkin Research, Greenwood Village, Colorado
  - Skin Research Institute, Coral Gables, Florida
  - Grekin Skin Institute, Warren, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Mercy Research, Washington, Missouri
  - Skin Specialists, PC, Omaha, Nebraska
  - Juva Skin & Laser Center, New York, New York
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Westlake Dermatology Clinical Research Center, Austin, Texas

IPD SHARING:
Plan to Share IPD: No